CLINICAL TRIAL: NCT04875182
Title: The Relationship Between Zonulin and Interleukin-8 Levels and Postoperative Delirium Development in Patients Who Had Femur Fracture Surgery Under Regional Anesthesia
Brief Title: The Relationship Between Zonulin and Interleukin-8 Levels and Postoperative Delirium Development
Acronym: ZolDel
Status: Completed | Type: Observational
Sponsor: Dr. Gokhan Vural (Other)
Responsible Party: Sponsor-Investigator, Dr. Gokhan Vural, Anesthesiologist Dr. Gokhan, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Other Study IDs: 26.02.2020- 04/VI
Record Dates: First submitted 2021-04-30; First posted 2021-05-06 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group delirium: Patients who are over 65 years of age and scheduled for femur fixation surgery will be included in the study. Blood samples for zonulin and interleukin-8 levels will be taken at the day prior to the surgery. All patients will be evaluated by Delirium Rating Scale for delirium development at the postoperative 1., 2. and 3. days. Patients with a Delirium Rating Scale-Revised-98 score of 11 points or higher will be included in the Group Delirium. And second blood samples for zonulin and interleukin-8 levels will be taken at the time of diagnosis.
  Postoperative pain scores of the patients will recorded by using a numerical rating scale.
  Interventions: Diagnostic Test: Evaluation of Delirium development
- group control: Patients who are over 65 years of age and scheduled for femur fixation surgery will be included in the study. Blood samples for zonulin and interleukin-8 levels will be taken at the day prior to the surgery. All patients will be evaluated by Delirium Rating Scale for delirium development at the postoperative 1., 2. and 3. days. Patients with a Delirium Rating Scale-Revised-98 score under 11 points for postoperative 72 hours will be included in the Group Control. And second blood samples for zonulin and interleukin-8 levels will be taken at the postoperative 72. hour.
  Postoperative pain scores of the patients will recorded by using a numerical rating scale.
  Interventions: Diagnostic Test: Evaluation of Delirium development

INTERVENTIONS:
Diagnostic Test: Evaluation of Delirium development — Postoperative pain scores of the patients will recorded by using a numerical rating scale.
  Other Names: Postoperative pain evaluation

SUMMARY:
The relationship between zonulin and interleukin-8 levels and postoperative delirium development in patients who had femur fracture surgery under regional anesthesia

DETAILED DESCRIPTION:
Patients who are over 65 years of age and scheduled for femur fixation surgery will be included in the study. Blood samples for zonulin and interleukin-8 levels will be taken at the day prior to the surgery. All patients will be evaluated by the Turkish version of the Delirium Rating Scale-Revised-98 (DRS-R-98) for delirium development at the postoperative 1., 2. and 3. days. Patients with a DRS-R-98 score of 11 points or higher will be included in the Group Delirium. And second blood samples for zonulin and interleukin-8 levels will be taken at the time of diagnosis.

Postoperative pain scores of the patients will recorded by using a numerical rating scale (NRS).

ELIGIBILITY:
Inclusion Criteria:

* patients over 65 years with mini mental state score > 21, undergoing femur fixation surgery

Exclusion Criteria:

* anticholinergic drug use, known epilepsy, Parkinson, Alzheimer's disease, dementia, cognitive function disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Both male and female patients over 65 years of age who will undergo femur neck and inthertrocanteric fracture surgery with regional anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
preoperative Zonulin | in the preoperative 24. hour
  The relation between postoperative delirium development and preoperative blood zonulin levels. The correlation between them will be analyzed by statistical analysis.
postoperative Zonulin | At the postoperative 72. hour
  The relation between postoperative delirium development and postoperative blood zonulin levels The correlation between them will be analyzed by statistical analysis.

SECONDARY OUTCOMES:
preoperative Interleukin-8 | in the preoperative 24. hour
  The relation between postoperative delirium development and preoperative blood interleukin-8 levels. The correlation between them will be analyzed by statistical analysis.
postoperative Interleukin-8 | At the postoperative 72. hour
  The relation between postoperative delirium development and postoperative blood interleukin-8 levels. The correlation between them will be analyzed by statistical analysis.

OTHER OUTCOMES:
Postoperative pain | At the postoperative 0., 12., 24 hours
  The relation between postoperative delirium development and postoperative pain score will be documanted. the scores are; zero; have no pain. 0-4 points: mid pain. 5-7points: mild pain. 8-10 points pain score will be named severe pain scores. and The correlation between them will be analyzed by statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan vural, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Sıtkı Koçman University, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no IPD will be shared with other researchers or anyone else